CLINICAL TRIAL: NCT00566813
Title: Islet Transplantation in Type 1 Diabetic Patients Using the Edmonton Protocol of Steroid Free Immunosuppression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jose Oberholzer, Professor, Division of Transplantation, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND11807-2004-0532
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Islets of Langerhans Transplantation; Exenatide; Soluble tumor necrosis factor receptor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation; Etanercept; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Islet Cell Transplant) (Active Comparator): 1-3 Islet transplants by the Edmonton Protocol of Steroid Free Immunosuppression using daclizumab 1 mg/kg IV immediately pre-transplant and 2, 4, 6, and 8 weeks after transplant; sirolimus dosed to maintain serum trough levels 12-15 ng/mL for three months post-transplant and 7-10 ng/mL therafter; tacrolimus dosed to maintain serum trough levels 3-6 ng/mL throughout the study.
  Interventions: Drug: Islet Cell Transplant
- Group 2 (Islet Cell Transplant plus) (Active Comparator): 1-3 islet transplants by the Edmonton Protocol of Steroid Free Immunosuppression using daclizumab 1 mg/kg IV immediately pre-transplant and 2, 4, 6, and 8 weeks after transplant; sirolimus dosed to maintain serum trough levels 12-15 ng/mL for 3 months post-transplant and 7-10 mg/mL thereafter; tacrolimus dosed to serum trough levels 3-6 ng/mL throughout the study; etanercept 50 mg IV pre-transplant, 25 mg subcutaneously post-transplant Days 3, 7, 10; exenatide 5-mcg subcutaneously twice daily for I week, then up to 10-mcg twice daily for 6 months after the last islet transplant.
  Interventions: Drug: Islet Cell Transplant plus

INTERVENTIONS:
Drug: Islet Cell Transplant — 1-3 allogeneic islet transplants; two doses of basiliximab 20 mg iv.; sirolimus po trough levels 10-15 ng/ml X 3 months, then 7-10 ng/ml; tacrolimus po trough levels 3-6 ng/ml
  Other Names: Allogeneic islets
  Arms: Group 1 (Islet Cell Transplant)
Drug: Islet Cell Transplant plus — 1-3 allogeneic Islets of Langerhans transplantations; two doses of basiliximab 20 mg iv.; sirolimus po daily to maintatin serum levels 12-15 ng/mL for 3 months, and 7-10 ng/mL thereafter; tacrolimus po twice daily to maintain serum levels 3-6 ng/mL; etanercept 50 mg IV before islet transplant, 25 mg subcutaneously post-transplant days 3, 7, 10; exenatide subcutaneously 5 mcg pre-transplant and twice daily for I week, then increased to 10-mcg twice daily for 6 months after the last islet transplant.
  Other Names: Islet Cell Transplant + Etanercept + Exenatide
  Arms: Group 2 (Islet Cell Transplant plus)

SUMMARY:
The primary purpose of this study is to demonstrate the safety of allogeneic islet transplantation in type 1 diabetic patients performed at the University of Illinois at Chicago (UIC). The purpose is to reproduce the Edmonton protocol to demonstrate that pancreatic islets isolated at UIC are safe and of sufficient quality to provide reproducible graft function.

DETAILED DESCRIPTION:
Diabetes mellitus is becoming an unbearable burden for the health care system worldwide. The incidence of disease has increased over the past 50 years, both for type I and type II diabetes. In 2002, the expenditure for direct and indirect costs of diabetes reached the astronomical amount of $132 billion for the USA alone. The burden suffered by patients is also grave when we consider that diabetic neuropathy and retinopathy are now the leading causes of renal failure and blindness in industrialized countries. Although major improvements in insulin treatment and glycemic control have been achieved, the development of hypoglycemic unawareness still represents a challenging clinical problem in the management of diabetes. Severe hypoglycemic episodes are not only acutely life threatening but lead to overall impairment of the quality of life of diabetic patients. Even under ideal study conditions the pathophysiology of hypoglycemic unawareness is not fully understood. It seems that each hypoglycemic episode reduces the counterregulatory hormone responses and the subjective awareness of the following episode, generating a self-worsening mechanism. Islet transplantation can effectively eliminate severe hypoglycemia and restore good glycemic control. However, there are still several limitations to the widespread application of islet transplantation. First, insulin independence is mostly achieved by transplanting a high number of islets that are harvested from 2-4 donors. Second, post-transplant insulin-independence is progressively lost over time despite continued endogenous insulin secretion. Lastly, current immunosuppression carries potential risks and can only incompletely prevent sensitization of the host and rejection.

At present, clinical trials in islet transplantation face stringent federal regulations, which define islets as a biological drug and islet transplantation as an experimental procedure. Limited resources impose small and uncontrolled trials investigating a limited number of new interventions to improve outcomes.

This study is a Phase 1/2 single center, uncontrolled trial in which 1-3 allogeneic pancreatic islet transplants are performed for each study subject. Post-transplant follow-up continues for 64 weeks after the final islet transplantation. Thereafter, subjects are enrolled for a 5-year follow-up study and a 5 to 10 year follow-up study.

The safety of islet transplantation depends primarily on the incidence of serious and unexpected complications or adverse events and the ability of the cell isolation laboratory to produce uncontaminated islet cell preparations with minimal endotoxin content. All study subjects are followed for safety for one year. An independent Data Monitoring Committee (DMC), composed of 3 members who have training in medicine and/or organ transplantation, will review eligibility and safety data approximately 2 weeks after each islet transplantation and every two months thereafter. An independent monitor knowledge on Good Clinical Practice(GCP) guidelines and regulations monitors the study for compliance with 21 CFR and according to ICH GCP Guidelines. Within the Clinical Research Center, the Scientific Advisory Committee and the Research Subject Advocacy Program monitor safety. These entities report to the Institutional Review Board, which also reviews safety data annually and on occurrence of serious adverse events. The principal investigator also report serious adverse events to the US Food and Drug Administration (FDA).

Success: Islet transplantation is considered a success when subjects do not use insulin and they achieve a fasting glucose level not exceeding 140 mg/dL more than three times in a week, and not exceeding two-hour post-prandial values of 180 mg/dL more than four times in a week.

Partial Success: Subjects who have a reduction in insulin requirements but who do not achieve insulin independence and present with a reduction in HbA1c and number of hypoglycemic episodes are considered to have partial success of islet transplantation. Reduction in insulin-requirements are assessed by comparing the pre-transplant insulin requirement recorded over two consecutive days (expressed as insulin units per kg) with the requirement on the two consecutive days preceding the subsequent islet infusion, and the requirements on two consecutive days at six months and again on two consecutive days at one year after the final transplant.

Failure: Absence of measurable levels of C-peptide after transplantation is considered as failure of islet cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes > 5 years complicated by at least one of the following situations despite intensive insulin management:

  * Reduced awareness of hypoglycemia at plasma glucose levels < 54 mg/dL
  * Metabolic lability/instability characterized by two or more episodes of severe hypoglycemia or hospital visits for diabetic ketoacidosis over the last year
  * Progressive secondary complications of diabetes:

    * Retinopathy-three step progression using the ETDRS grading system or equivalent progression;
    * Nephropathy- microalbuminuria rise of 50 µg/min (72 mg/24h) over three months within the past two years despite using an ACE inhibitor;
    * Neuropathy-persistent gastroparesis, postural hypotension, neuropathic bowel or bladder, or severe peripheral neuropathy unresponsive to management

Exclusion Criteria:

* Co-existing cardiac disease:

  * Myocardial infarction within past six months
  * Angiographic evidence of non-correctable coronary artery disease
  * Ischemia on functional cardiac exam d. Heart failure > NYHA II
* Active alcohol or substance abuse or cigarette smoking
* Psychiatric disorder: schizophrenia, bipolar disorder, or major depression that is unstable on medication
* Non-adherence to prescribed regimens
* Active infection including hepatitis C, hepatitis B, HIV
* TB by history, current infection, or under treatment for suspected TB
* History of malignancies except squamous or basal skin cancer
* Stroke within the past 6 months
* BMI > 26 kg/m2 or body weight > 70 kg at screening visit
* C-peptide response to glucagon stimulation, any C-peptide ≥ 0.3 ng/mL
* Inability to provide informed consent
* Age less than 18 or greater than 65 years
* Creatinine clearance < 85 mL/min/1.73 m2 by 24-hour urine collection
* Serum creatinine > 1.5 mg/dL
* Macroalbuminuria > 300 mg/24h
* Baseline Hb < 12 gm/dL in women, < 13 gm/dL in men
* Baseline liver function tests outside normal range
* Untreated proliferative retinopathy
* Positive pregnancy test, intent for pregnancy, male's intent to procreate, unwilling to use effective contraception, breast-feeding
* Previous transplant or PRA reactivity > 20%)
* Insulin requirement > 0.7 IU/kg/day
* HbA1C > 12%
* Hyperlipidemia
* Chronic use of steroids
* Use of coumadin or other anticoagulant (except aspirin) or PT INR > 1.5
* Addison's disease
* Allergy to radiographic contrast material

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-11; Primary Completion 2010-07-05 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Oberholzer, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gangemi A, Salehi P, Hatipoglu B, Martellotto J, Barbaro B, Kuechle JB, Qi M, Wang Y, Pallan P, Owens C, Bui J, West D, Kaplan B, Benedetti E, Oberholzer J. Islet transplantation for brittle type 1 diabetes: the UIC protocol. Am J Transplant. 2008 Jun;8(6):1250-61. doi: 10.1111/j.1600-6143.2008.02234.x. Epub 2008 Apr 29. PMID 18444920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of adults ages 18-65 occurred from 10/22/2004 to 2/21/2006 when the 10th eligible participant was confirmed. Potential participants were recruited from physician referrals at University of Illinois (UIC) or private practice, from information posted on the UIC Transplant Division website, and from diabetes chat groups.
Pre-assignment Details: 88 individuals completed phone screenings; 15 withdrew, 58 excluded mainly for high weight, kidney disease, high insulin use, lack of hypoglycemia unawareness, previous transplant. 36 enrolled to be screened for eligibility. Of the 36, 5 withdrew, 21 were excluded for not meeting eligibility requirements. Remaining 10 subjects received transplants.
Groups:
- Group 1 (Islet Cells): 1-3 Islet transplants by the Edmonton Protocol of Steroid Free Immunosuppression using daclizumab 1 mg/kg IV immediately pre-transplant and 2, 4, 6, and 8 weeks after transplant; sirolimus dosed to maintain serum trough levels 12-15 ng/mL for three months post-transplant and 7-10 ng/mL therafter; tacrolimus dosed to maintain serum trough levels 3-6 ng/mL throughout the study.
- Group 2 (Islet Cells + Etanercept + Exenatide): 1-3 islet transplants by the Edmonton Protocol of Steroid Free Immunosuppression using daclizumab 1 mg/kg IV immediately pre-transplant and 2, 4, 6, and 8 weeks after transplant; sirolimus dosed to maintain serum trough levels 12-15 ng/mL for 3 months post-transplant and 7-10 mg/mL thereafter; tacrolimus dosed to serum trough levels 3-6 ng/mL throughout the study; etanercept 50 mg IV pre-transplant, 25 mg subcutaneously post-transplant Days 3, 7, 10; exenatide 5-mcg subcutaneously twice daily for I week, then up to 10-mcg twice daily for 6 months after the last islet transplant.
Period: Overall Study
Arm/Group | Group 1 (Islet Cells) | Group 2 (Islet Cells + Etanercept + Exenatide)
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Islet Cells: Islet transplantation and the Edmonton protocol of steroid free immunosuppression
- Islet Cells + Etanercept + Exenatide: Edmonton Protocol, etanercept ,exenatide
- Total: Total of all reporting groups
Arm/Group | Islet Cells | Islet Cells + Etanercept + Exenatide | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.9) | 44.5 (9.7) | 46.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Including Laboratory Abnormalities at the End of Study Participation
Description: * Frequency of adverse events including laboratory abnormalities
  * HbA1C (less than 6.1% is considered normal)
  * Glucose control and absence of hypoglycemic coma/unawareness, as evidenced by no further requirement for third-party assistance or hospital attendance resulting from a severe hypoglycemic episode
  * Renal function, measured both by serum creatinine and calculated GFR using the Cockroft & Gault
  * Lipid profiles for cholesterol, triglycerides, low density lipoprotein (LDL) and high density lipoprotein (HDL)
  * PRA
  * Doppler ultrasound to exclude or document portal vein thrombosis
  * Immunosuppressive drug trough levels
  * Renal clearance (GFR)
  * Liver function tests
  * Diagnosis of opportunistic infections, e.g., CMV
Time Frame: 15 months after the last transplant
Population: The number of participants analyzed represents the number of subjects in Group 1 (Islet Cells) and Group 2 (Islet Cells + Etanercept + Exenatide)
Measure: Number; unit: participants
Groups:
- Islet Cells: 1-3 Islet transplants by the Edmonton Protocol of Steroid Free Immunosuppression using daclizumab 1 mg/kg IV immediately pre-transplant and 2, 4, 6, and 8 weeks after transplant; sirolimus dosed to maintain serum trough levels 12-15 ng/mL for three months post-transplant and 7-10 ng/mL therafter; tacrolimus dosed to maintain serum trough levels 3-6 ng/mL throughout the study.
- Islet Cells + Etanercept + Exenatide: 1-3 islet transplants by the Edmonton Protocol of Steroid Free Immunosuppression using daclizumab 1 mg/kg IV immediately pre-transplant and 2, 4, 6, and 8 weeks after transplant; sirolimus dosed to maintain serum trough levels 12-15 ng/mL for 3 months post-transplant and 7-10 mg/mL thereafter; tacrolimus dosed to serum trough levels 3-6 ng/mL throughout the study; etanercept 50 mg IV pre-transplant, 25 mg subcutaneously post-transplant Days 3, 7, 10; exenatide 5-mcg subcutaneously twice daily for I week, then up to 10-mcg twice daily for 6 months after the last islet transplant.
Arm/Group | Islet Cells | Islet Cells + Etanercept + Exenatide
Number analyzed (Participants) | 4 | 6
participants | 4 | 5

2. Primary Outcome: Number of Participants With Insulin Independence at End of Study Participation
Description: Primary efficacy outcome: independence from insulin injections with adequate control of blood glucose in subjects with Type 1 diabetes. Transplant is considered a success when 2 weeks after their last transplant, subjects are not using insulin, and fasting glucose levels do not exceed 7.8 mmol/L (140 mg/dL) more than 3 times/week, and two-hour post-prandial glucose values do not exceed 10 mmol/L (180 mg/dL) more than 4 times/week. During the 15 months after last transplant, a subject will be considered a success if an illness or other event (e.g., high tacrolimus level) causes need for insulin not exceeding 14 days providing evidence of graft rejection is not apparent. The proportion of subjects who are insulin independent and meet criteria for glucose control will be determined at 2 weeks and 1, 3, 6, 12, and 15 months following their final islet transplant.
Time Frame: End of 15 Month Study Participation/Follow-up
Measure: Number; unit: participants
Arm/Group | Islet Cells | Islet Cells + Etanercept + Exenatide
Number analyzed (Participants) | 4 | 6
participants | 4 | 5

3. Primary Outcome: Number of Participants With HbA1c Less Than or Equal to 6.5 & Free of Severe Hypoglycemic Events
Description: HbA1c less than or equal to 6.5 at end of 15 month study participation, and lack of or free from severe hypoglycemic events, defined as an event with symptoms compatible with hypoglycemia in which the subject required the assistance of another person and which was associated with either a blood glucose level < 50 mg/dl (2.8 mmol/L) or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration.
Time Frame: At end of 15 month study participation
Measure: Number; unit: participants
Arm/Group | Islet Cells | Islet Cells + Etanercept + Exenatide
Number analyzed (Participants) | 4 | 6
participants | 4 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year following the last transplant.
Description: Review of Systems and adverse events at each study visit, physical examinations, notification from subjects.
Arm/Group | Islet Cells | Islet Cells + Etanercept + Exenatide
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Islet Cells (N=4) | Islet Cells + Etanercept + Exenatide (N=6)
Intrahepatic hematoma (Injury, poisoning and procedural complications) | 0 | 1
Intraperitoneal hematoma (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Cells (N=4) | Islet Cells + Etanercept + Exenatide (N=6)
Transient anemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Increased creatinine (Renal and urinary disorders) | 1 (1) | 2 (2)
Temporary nausea, vomiting, and weight loss (Gastrointestinal disorders) | 0 (0) | 6 (6) — Due to exenatide.
Scalene muscle myonecrosis and vertebral osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) — Due to staph aureus.
Irregular menstrual bleeding and ruptured ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Related to immunosuppressive medications. Treated with abdominal hysterectomy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No